CLINICAL TRIAL: NCT04723043
Title: The Effect of Pressure Controlled and Volume Controlled Ventilation Modes on Cerebral Oxymetry and Blood Gases In Laparoscopic Cholecystectomy Operations
Brief Title: The Effect of Ventilation Modes on Cerebral Oxymetry In Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emre Badur MD, specialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1305
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Cholecystitis; Gallstone; Mechanical Ventilation Pressure High; Intraabdominal Hypertension
Keywords: laparoscopy
MeSH Terms: conditions — Cholecystitis; Gallstones; Intra-Abdominal Hypertension

STUDY DESIGN:
Intervention Model Description: The first group was labelled as "Group V" as they are applied with mechanical ventilation under controlled volume, and the second group was labelled as "Group P" as they are applied with mechanical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- v group (Active Comparator): patients will ventilate with volume controlled mode
  Interventions: Device: mechanical ventilation modes
- p group (Active Comparator): patients will ventilate with pressure controlled mode
  Interventions: Device: mechanical ventilation modes

INTERVENTIONS:
Device: mechanical ventilation modes — ventilation with pressure controlled mode in laparoscopic abdominal surgery ventilation with volume controlled mode in laparoscopic abdominal surgery

SUMMARY:
In laparoscopic cholecystectomy method, Insufflation of CO2 in abdominal cavity causes positioning of the diaphragm upwards, a decrease in lung's volume and its compliance, an increase in the airway resistance, mismatch between the atelectasis and the ventilation perfusion. Although there are numerous studies in laparoscopic surgery, only a few of them investigate the effects of laparoscopic surgery on the cardiopulmonary and the respiratory mechanics. The investigator aimed To examine the effects of pressure-controlled and volume-controlled ventilation modes on cerebral oximetry and blood gases in laparoscopic cholecystectomy operations.

DETAILED DESCRIPTION:
Since the laparoscopic methods have been introduced to the surgical operations, laparoscopic cholecystectomy has become the golden standard in gall bladder surgical treatments. In this method, carbon dioxide (CO2) pneumoperitoneum method is used to achieve the desired surgical and visual conditions. Alongside the advantages of the Laparoscopic cholecystectomy method (e.g. shortening the patient's length of stay at the hospital, minimal postoperative pain and rapid recovery), it has various intraabdominal pressure related systemic disadvantages . Insufflation of CO2 in abdominal cavity causes positioning of the diaphragm upwards, a decrease in lung's volume and its compliance, an increase in the airway resistance, mismatch between the atelectasis and the ventilation perfusion. Various ventilation strategies have been introduced to increase arterial oxygenation, functional residual capacity (FRC), and the lung compliance. Recent studies; demonstrates that pressure-controlled mechanical ventilation is superior to volume-controlled mechanical ventilation in providing arterial and tissue oxygenation.

Although there are numerous studies in laparoscopic surgery, only a few of them investigate the effects of laparoscopic surgery on the cardiopulmonary and the respiratory mechanics. Several experimental and clinical studies describe that the cardiovascular effects of the high intraabdominal pressure and the CO2 insufflation is complex. In fact, the results are linked to the studied patients' population, the lung's position and its volume. As it is known in laparoscopic surgeries, the oxygenation in cerebral tissue decreases as the intraabdominal pressure increases. At present, bispectral index (BIS), electroencephalography (EEG), auditory evoke potential (AEP) (and several others) and functional NIRS (fNIRS) are used to measure cerebral oxygenation and anaesthetic depth. NIRS monitorisation makes use of the combined effects of the transmission, the reflection, the dispersion, and the absorption of light. It can also measure the oxygen saturation in tissues that does not have pulsatile circulation. The investigator aimed To examine the effects of pressure-controlled and volume-controlled ventilation modes on cerebral oximetry and blood gases in laparoscopic cholecystectomy operations.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology) score of 1 and 2
* body mass index < 30 kg/m2
* planned elective laparoscopic cholecystectomy operation
* 18-65 years old

Exclusion Criteria:

* who are applied with emergency laparoscopic cholecystectomy operation
* ASA (American Society of Anesthesiology) score of 3 and above
* hematocrit value 30 and below
* body mass index> 30 kg/m2
* major pulmonary disease (this condition was defined as having capacity and currency flow speed values that are below %70 in respiratory functional tests)
* patients with a history of thoracic surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
NIRS | 0 to 3 hours (approximately)
  near infrared reflectance spectroscopy values recorded at before the anesthesia, after intubation, before and after deflation
oxygen saturation | 0 to 3 hours (approximately)
  oxygen saturation with pulse-oximeter at before the anesthesia, after intubation, before and after deflation
end-tidal carbon dioxide | 0 to 3 hours (approximately)
  end-tidal carbon dioxide with mechanical ventilator at before the anesthesia, after intubation, before and after deflation

SECONDARY OUTCOMES:
partial oxygen pressure | 0 to 3 hours (approximately)
  partial oxygen pressure in blood gases at before the anesthesia, after intubation, before and after deflation
P peak | 0 to 3 hours (approximately)
  peak pressure in mechanical ventilation mod at before the anesthesia, after intubation, before and after deflation

CONTACTS AND LOCATIONS:
Overall Officials: ayse surhan cinar, Study Director — chief of anesthesia department
Locations (1):
- Sisli Etfal Research and Training Hospital, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gipson CL, Johnson GA, Fisher R, Stewart A, Giles G, Johnson JO, Tobias JD. Changes in cerebral oximetry during peritoneal insufflation for laparoscopic procedures. J Minim Access Surg. 2006 Jun;2(2):67-72. doi: 10.4103/0972-9941.26651. PMID 21170237
- [Background] Casati A, Fanelli G, Pietropaoli P, Proietti R, Tufano R, Danelli G, Fierro G, De Cosmo G, Servillo G; Collaborative Italian Study Group on Anesthesia in Elderly Patients. Continuous monitoring of cerebral oxygen saturation in elderly patients undergoing major abdominal surgery minimizes brain exposure to potential hypoxia. Anesth Analg. 2005 Sep;101(3):740-747. doi: 10.1213/01.ane.0000166974.96219.cd. PMID 16115985
- [Background] Nielsen HB. Systematic review of near-infrared spectroscopy determined cerebral oxygenation during non-cardiac surgery. Front Physiol. 2014 Mar 17;5:93. doi: 10.3389/fphys.2014.00093. eCollection 2014. PMID 24672486